CLINICAL TRIAL: NCT02095834
Title: A Single Center Phase Ib Study of Carfilzomib, Bendamustine, and Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Carfilzomib, Bendamustine Hydrochloride, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0162; NCI-2014-00884 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0162 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dexamethasone, bendamustine, carfilzomib) (Experimental): Patients receive dexamethasone PO or IV over 20 minutes on days 1, 2, 8, 9, 15, 16, 22, and 23 of courses 1-3; on days 1, 2, 15, and 16 of courses 4-12; and on days 1 and 2 of all subsequent courses. Patients also receive bendamustine hydrochloride IV over 10 minutes on days 1 and 2 of courses 1-3 and on day 1 of all subsequent courses and carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16 of courses 1-12 and on days 1, 2, 15, and 16 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Carfilzomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase Ib trial studies the side effects and best doses of carfilzomib and bendamustine hydrochloride when given together with dexamethasone in treating patients with multiple myeloma that has returned or does not respond to treatment. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as bendamustine hydrochloride, work to stop the growth of cancer cells by killing the cells. Biological therapies, such as dexamethasone, may stimulate the immune system and stop cancer cells from growing. Giving carfilzomib, bendamustine hydrochloride, and dexamethasone may be a better way to treat multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of carfilzomib in combination with bendamustine (bendamustine hydrochloride) and dexamethasone, up to a maximum bendamustine dose of 90 mg/m^2.

SECONDARY OBJECTIVES:

I. To evaluate the safety of carfilzomib in combination with bendamustine and dexamethasone, at the MTD.

II. To evaluate the response rate and duration of response of carfilzomib in combination with bendamustine and dexamethasone, in patients with relapsed and or refractory multiple myeloma.

OUTLINE: This is a dose-escalation study of carfilzomib and bendamustine hydrochloride.

Patients receive dexamethasone orally (PO) or intravenously (IV) over 20 minutes on days 1, 2, 8, 9, 15, 16, 22, and 23 of courses 1-3; on days 1, 2, 15, and 16 of courses 4-12; and on days 1 and 2 of all subsequent courses. Patients also receive bendamustine hydrochloride IV over 10 minutes on days 1 and 2 of courses 1-3 and on day 1 of all subsequent courses and carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16 of courses 1-12 and on days 1, 2, 15, and 16 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and or refractory multiple myeloma after at least one prior line of therapy; there is no upper limit of prior lines of therapy; patients who are ineligible for stem cell transplantation are allowed; patients should have received at least one prior novel agent (immunomodulatory agents or proteasome inhibitors); patients eligible for bone marrow transplant must have undergone bone marrow transplant (BMT) prior to enrollment
* Measurable disease, as defined by one or all of the following (assessed within 30 days prior to initiation of therapy): a) serum M-protein >= 0.5 g/d; b) urine Bence-Jones protein >= 200 mg/24 hours; c) patients with light chain only myeloma are eligible; the involved free light chain level 100 mg/L with abnormal serum free light chain ratio
* Documented relapse or progressive disease on or after any regimen (subjects refractory to the most recent regimen are eligible)
* Primary refractory patients (never responded to any therapy) are eligible
* Eastern Cooperative Oncology Group performance status 0 - 2
* Serum alanine aminotransferase (ALT) < 3.5 times the upper limit of normal within 30 days prior to cycle 1 day 1
* Serum direct bilirubin < 2 mg/dL (34 Omol/L) within 30 days prior to cycle 1 day 1
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L within 30 days prior to cycle 1 day 1, without granulocyte-colony stimulating factor (G-CSF)
* Hemoglobin > 9 g/dL (80 g/L) within 30 days prior to cycle 1 day 1 (subjects may be receiving red blood cell transfusions in accordance with institutional guidelines)
* Platelet count > 100 x 10^9/L (30 x 10^9/L if myeloma involvement in the bone marrow aspirate is > 50%) within 30 days prior to cycle 1 day 1; subjects may receive platelet transfusions within institutional guidelines
* Creatinine clearance > 50 mL/minute within 30 days prior to cycle 1 day 1, either measured or calculated using a standard formula
* Patient should have a normalized or normal uric acid level prior to study entry
* Written informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential must have a negative pregnancy test and agree to ongoing pregnancy testing and to practice contraception; (birth control methods should be determined in consultation with the investigator)
* Male subjects must agree to practice contraception

Exclusion Criteria:

* Intolerance to previous bendamustine, carfilzomib or dexamethasone or mannitol; subjects who are allergic to bortezomib are not excluded
* Chemotherapy (approved or investigational) within 3 weeks prior to the first day of treatment or antibody therapy within 6 weeks prior to the first day of treatment
* Radiotherapy to >= 3 sites at the same time within 1 week prior to the first day of treatment
* Immunomodulatory therapy such as immunomodulatory drugs (Imids) or stem cell transplant within 28 days prior to the first day of treatment
* Pregnant or lactating females
* Major surgery within 21 days prior to the first day of treatment
* Acute active infection requiring treatment (IV antibiotics, antivirals, or antifungals) within 14 days prior to the first day of treatment
* Known human immunodeficiency virus infection
* Known active hepatitis B or C infection
* Unstable angina or myocardial infarction within 4 months prior to the first day of treatment, the New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or grade 3 conduction system abnormalities unless subject has a pacemaker
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to the first day of treatment
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (grades 3 - 4, or grade 2 with pain) within 14 days prior to the first day of treatment
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Subjects with known or likely systemic amyloidosis
* Ongoing graft-vs-host disease
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to the first day of treatment
* Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of carfilzomib and bendamustine hydrochloride when given together with dexamethasone, defined as the dose level below which dose limiting toxicity is observed in greater than or equal to 33% of subjects | 28 days
Recommended Phase 1b dose of carfilzomib and bendamustine hydrochloride when given together with dexamethasone | Up to 6 years
  The Phase 1b recommended dose of both agents will be determined from a qualitative assessment of a broad set of considerations that include the following: safety and tolerability, disease response, and biologic activity.

SECONDARY OUTCOMES:
Best overall response, including stringent complete remission, complete remission, very good partial remission, and partial remission | 112 days (4 courses of therapy)
  Overall response will be defined using the International Myeloma Working Group Uniform Response Criteria, with the addition of minimal response according to the European Group for Blood and Marrow Transplant criteria.

OTHER OUTCOMES:
Duration of objective response | Up to 6 years
Progression free survival | Up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org